CLINICAL TRIAL: NCT01999140
Title: Implantable Cardioverter Defibrillator (ICD Registry)
Status: Recruiting | Type: Observational
Sponsor: American College of Cardiology (Other)
Responsible Party: Sponsor
Other Study IDs: ICD Registry
Record Dates: First submitted 2013-11-19; First posted 2013-12-03 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure; Nonischemic Cardiomyopathy; Ischemic Cardiomyopathy; Ventricular Arrhythmia; Complications; Device, Cardiac
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Primary prevention

SUMMARY:
The ICD Registry™ is a nationwide quality program that helps participating hospitals measure and improve care for patients receiving implantable cardioverter defibrillators (ICDs) and cardiac resynchronization therapy devices with defibrillator (CRT-Ds). The ICD Registry captures the characteristics, treatments, and outcomes of patients receiving (ICDs). Patient-level data is submitted by participating hospitals on a quarterly basis to the American College of Cardiology Foundation's (ACCF) National Cardiovascular Data Registry (NCDR) which then produces an Outcomes Report of the hospital's data, with comparison to both a volume peer group (number of ICD patients submitted annually) and the entire ICD registry data set.

DETAILED DESCRIPTION:
In January 2005 the Centers for Medicare and Medicaid Services (CMS) expanded the covered indications for primary prevention implantable cardioverter defibrillators (ICDs) to incorporate the findings from the Sudden Cardiac Death Heart Failure Trial (SCDHeFT) and the Multicenter Automatic Defibrillator Implantation Trial II (MADIT II). As part of this expansion, CMS mandated that a national registry be formed to compile data on Medicare patients implanted with primary prevention ICDs to confirm the appropriateness of ICD utilization in this patient population.

Responding to this mandate, a collaborative effort of the Heart Rhythm Society (HRS)and the American College of Cardiology Foundation (ACCF), utilizing the expertise of the National Cardiovascular Data Registry (NCDR®), developed the ICD Registry™. Enrollment opened on June 1, 2005. CMS selected the NCDR ICD Registry as the mandated national registry in October 2005.

ELIGIBILITY:
All U.S and International patients.

Inclusion Criteria:

* All patients who receive an ICD/CRT-D (initial or generator change) for primary or secondary prevention purposes.
* All patients with an ICD/CRT-D undergoing a Lead Only procedure.
* U.S. populations must submit all patients who receive an ICD/CRT-D (initial or generator change) for primary prevention purposes who are insured by Medicare.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All facilities performing ICD implants
Sampling Method: Non-Probability Sample
Enrollment: 1750 (Estimated)
Dates: Start 2005-06; Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Risk Adjusted Complications and Death Composite Measure | Post-procedure until discharge occurences. Reported quarterly based on a rolling 1 year of data.
  Reported as one value for a composite measure looking at the following complications and death: Cardiac arrest, cardiac perforation, coronary venous dissection, hemothorax, device-related infection, lead dislodgement, mortality, myocardial infarction, pericardial tamponade, pneumothorax, stroke/transischemic attack (TIA), urgent cardiac surgery, hematoma, set screw problem

CONTACTS AND LOCATIONS:
Locations (1):
- American College of Cardiology/National Cardiovascular Data Registry (NCDR), Washington D.C., District of Columbia, United States

REFERENCES:
- See also: The link will provide further information about the ICD Registry as well as related research and publications. — https://www.ncdr.com/webncdr/icd/